CLINICAL TRIAL: NCT02072200
Title: A New Modified-Release Tablet Formulation of Prednisone in Patients With Rheumatoid Arthritis- Multicenter, Phase IV, Interventional Study to Assess Reduction of Morning Stiffness
Brief Title: Efficacy of Lodotra®(Prednisone) in Reduction of Morning Stiffness Duration(K-IMPROvE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOD13-KR-401
Record Dates: First submitted 2014-02-14; First posted 2014-02-26 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
Keywords: RA, MS, Safety, Efficacy, MR prednisone
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modified release prednisone (Experimental): Single arm / Lodotra
  Interventions: Drug: Lodotra®

INTERVENTIONS:
Drug: Lodotra® — Single arm will be received below oral 10mg tablet daily and maximum 10mg/d depending on the clinical symptoms and the patient's response
  Other Names: Modified Release Prednisone

SUMMARY:
This study is multicenter, Ph IV, single arm, interventional study to assess relative reduction of morning stiffness of Lodotra® in Rheumatoid Arthritis patients.Study medication will start after study visit at baseline (week 0, visit 1) and follow-up visit will be after 2, 6 and 12 weeks after treatment (visit 2,3,4).

DETAILED DESCRIPTION:
Test Treatment, Dose, and Mode of Administration:

Starting dose is 10mg, and depending on the clinical symptoms and the patient's response, the initial dose can quickly be reduced to a lower maintenance dose. When changing over from the standard regimen (glucocorticoid administration in the morning) to Lodotra® administered at bedtime (at about 10 pm), the same dose (in mg prednisone equivalent) should be maintained, if the subject has taken stable dose within 30 days. Lodotra® dose cannot exceed more than 10mg.

Lodotra® should be taken at bedtime (at about 10 pm), with or after the evening meal and be swallowed whole with sufficient liquid. If more than 2 - 3 hours have passed since the evening meal, it is recommended to take Lodotra® with a light meal or snack.

Modified-release tablets are not to be broken, divided or chewed.

Treatment procedure:At Visit 1(week 0), subjects who qualify for entry into the study will medicated to Lodotra® starting dose of 10 mg daily. (Written informed consent has to be obtained, and subjects will undergo complete evaluation for study eligibility) No dose increase will be allowed for more than 10mg

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed more than 3 months
* Morning stiffness on previous treatment with or without oral steroids (below or equal to 10mg per day, methylprednisolone doses were converted into prednisone doses as follows: prednisone dosed=methylprednisolone dose*1.25), average daily duration of 45 min or more.
* Average daily maximum pain intensity score (100 mm VAS) of 30mm or more.
* DAS-ESR ≥3.2
* On DMARD treatment including MTX for ≥3months and stable treatment dose within the past 30 days. There are no limitations on number of DMARDs treatment.(Except patients who have experience of adverse drug reaction of MTX or difficulty to administer MTX due to disease specific condition.)
* Able to perform study procedures and given written informed consent.
* Naïve patients with Prednisone MR(Lodotra® ) or patients not treat with Prednisone MR(Lodotra®) within 4 weeks(28days)
* Subject who keeps to administer study drug at 22±30 daily
* Subject who provide signed and dated written voluntary informed consent

Exclusion Criteria:

* Patients who suffers from another disease, which requires glucocorticoid treatment during the study period.
* Synovectomy within 4 months prior to study start.
* Patients who underwent joint injections on only fingers and wrists(both sides) within 4 weeks prior to first visit. Clinically significant disease which, in the investigator's opinion, would exclude the subject from the study.
* Significant renal impairment (serum creatinine>2.0mg/dl)
* Significant hepatic impairment (>3 times the upper limit of normal range in each site)
* All contra-indications for glucocorticoids.(established new osteoporotic fractures history of corticoid psychosis, herpes simplex and herpes zoster, varicella infection)
* Uncontrolled DM(HbA1c>8.0)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant. UNLESS they are:

  * women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner
  * women whose partners have been sterilized by vasectomy or other means
  * two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test
* Participation in another clinical study within the past 30 days
* Known hypersensitivity to prednisone
* Infection patients without effective antimicrobial and systemic mycosis infection patients(infection might be aggravated due to suppression of immunologic function.)
* Patients with immunization with live vaccines within 2 weeks of enrollment or planned during the study
* Since this drug contains glucose, patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption should not take this drug.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seungjae Hong, PhD, Principal Investigator — Kyunghee University Hospital
Locations (1):
- Hallym University Sacred Heart Hospital, Pyeongchon, Kyungkido, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modified Release Prednisone
Started | 147
Completed | 145
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: These 145 subjects received at least 1 dose of study drug and completed the study.
Arm/Group | Modified Release Prednisone
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: participant] | 55.41 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 32
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 145

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Stiffness Duration at Week 12 as Assessed by Patient Diary
Description: Data for the duration of morning stiffness will be obtained from patient diaries. Duration of morning stiffness will be from wake-up time to time of resolution of morning stiffness.
  Relative reduction rate of the morning stiffness duration from baseline to Week 12 of the study drug treatment was calculated for this outcome measure.
Time Frame: Baseline and 12 weeks
Population: ITT set = 145 patients. Missing data was handled as LOCF.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Modified Release Prednisone
Number analyzed (Participants) | 145
minutes | -16.76 (3.352)

2. Secondary Outcome: Change of Baseline Severity of Morning Stiffness at Week 12 Using Visual Analog Scale (VAS) Scale
Description: The VAS is a 100 mm line ranging from 0 mm (no pain) on the left end and 100 mm (worst pain) on the right end. Subjects marked on the line to indicate their pain severity. The distance in mm was measured from the left end to the subject's marking.
Time Frame: Baseline and 12 weeks
Population: ITT population was 145, but 3 patients were not assessed for primary efficacy parameter of morning stiffness severity. So, Last Observation Carried Forward (LOCF) was not done for these 3 patients after baseline . Other patients' missing data were handled using LOCF method.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Modified Release Prednisone
Number analyzed (Participants) | 142
mm | -25.70 (25.87)

3. Secondary Outcome: Change of Functional Disability Index of the Korea Health Assessment Questionnaire (KHAQ) From Baseline to Week 12
Description: Change in KHAQ score from baseline to Week 12 post-treatment: KHAQ is composed of 8 functional disability indices. The scale for each index is from 0 (without any difficulty) to 3 (unable to do). Scores for each disability index were summed to obtain the total score for each subject, ranging between 0 to 24, with higher scores reflecting higher functional disability. The scores were then averaged across all subjects.
Time Frame: 12 weeks
Population: ITT set was 145 patients, but 11 patients data was not assessed except baseline score.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Modified Release Prednisone
Number analyzed (Participants) | 134
scores on a scale | -4.76 (8.16)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Modified Release Prednisone
Serious Adverse Events (participants affected / at risk) | 5/145
Other Adverse Events (participants affected / at risk) | 51/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Modified Release Prednisone (N=145)
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Modified Release Prednisone (N=145)
Nasopharyngitis (Infections and infestations) | 6
Dyspepsia (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea, vomiting, constipation, gastric disorder, gastritis, gastrointestinal disorder (Gastrointestinal disorders) | 8
Bronchitis, cellulitis, conjunctivitis, folliculitis, rhinitis (Infections and infestations) | 5
Joint swelling, musculoskeletal pain, neck pain, pain in extremity, synovial cyst (Musculoskeletal and connective tissue disorders) | 5
Face edema, edema, pain, pyrexia, oedma peripheral (General disorders) | 8
Alanine aminotransferase increased, aspartate aminotransferase increased, blood glucose increased (Investigations) | 3
Alopecia, onychoclasis, rash, urticaria (Skin and subcutaneous tissue disorders) | 4
Cataract, dry eye, eyelid edema, vision blurred (Eye disorders) | 4
Humerus fracture, thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2
Hyperlipedemia (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI/ Institution shall provide to Mundipharma any proposed presentation at least 15 working days prior to being disclosed and any other proposed publication at least 45 working days prior to being disclosed. Mundipharma may in its sole discretion permit such publications and presentations and shall have the right to require amendments to any such proposed presentation or publication on reasonable grounds.